CLINICAL TRIAL: NCT01451320
Title: Comparison of Different TRansesophageal Echocardiography Guided thrOmbolytic Regimens for prosthetIc vAlve Thrombosis
Acronym: TROIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, MEHMET OZKAN, Principal Investigator, MD., FESC., Assoc. Prof,. Head of Cardiology, Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11
Record Dates: First submitted 2011-09-29; First posted 2011-10-13 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Prosthetic Valve Thrombosis
Keywords: Prosthetic valve; thrombosis; TROIA; tPA; TEE
MeSH Terms: conditions — Thrombosis | interventions — Streptokinase; Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- rapid streptokinase (Active Comparator): 3-hour infusion of 1.5 million units of streptokinase (16 patients, 16 episodes), repeat once 24 hours later if needed (maximum total dose 3 million units).
  Interventions: Drug: Streptokinase
- high dose tpa (Active Comparator): 5-hour infusion of 90 mg t-PA(Tissue plasminogen activator) after 10 mg bolus (10 patients, 12 episodes), repeat once 24 hours later if needed (maximum total dose 200 mg)
  Interventions: Drug: Tissue plasminogen activator
- slow streptokinase (Active Comparator): 24-hour infusion of 1.5 million units of streptokinase (41 patients, 41 episodes), repeat once 24 hours later if needed (maximum total dose 3 million units).
  Interventions: Drug: Streptokinase
- half-dose slow infusion tpa (Active Comparator): 6-hour infusion of 50 mg t-PA (Tissue plasminogen activator) without bolus (27 patients, 27 episodes), repeat once 24 hours later up to 3 times if needed (maximum total dose 150 mg).
  Interventions: Drug: Tissue Plasminogen Activator
- low dose slow infusion tpa (Active Comparator): 6-hour infusion of 25 mg t-PA(Tissue plasminogen activator) without bolus (108 patients, 124 episodes), repeat once 24 hours later up to 6 times if needed (maximum total dose 150 mg).
  Interventions: Drug: Tissue Plasminogen Activator

INTERVENTIONS:
Drug: Streptokinase — 3-hour infusion of 1.5 million units of streptokinase (16 patients, 16 episodes), repeat once 24 hours later if needed (maximum total dose 3 million units)
  Other Names: Streptase
  Arms: rapid streptokinase
Drug: Streptokinase — 24-hour infusion of 1.5 million units of streptokinase (41 patients, 41 episodes), repeat once 24 hours later if needed (maximum total dose 3 million units).
  Other Names: Streptase
  Arms: slow streptokinase
Drug: Tissue plasminogen activator — 5-hour infusion of 90 mg t-PA (Tissue plasminogen activator) after 10 mg bolus (10 patients, 12 episodes), repeat once 24 hours later if needed (maximum total dose 200 mg)
  Other Names: ACTILYSE
  Arms: high dose tpa
Drug: Tissue Plasminogen Activator — 6-hour infusion of 50 mg t-PA (Tissue plasminogen activator) without bolus (27 patients, 27 episodes), repeat once 24 hours later up to 3 times if needed (maximum total dose 150 mg).
  Other Names: ACTILYSE
  Arms: half-dose slow infusion tpa
Drug: Tissue Plasminogen Activator — 6-hour infusion of 25 mg t-PA (Tissue plasminogen activator) without bolus (108 patients, 124 episodes), repeat once 24 hours later up to 6 times if needed (maximum total dose 150 mg).
  Other Names: ACTILYSE
  Arms: low dose slow infusion tpa

SUMMARY:
Despite high mortality and morbidity, the best treatment strategies for prosthetic valve thrombosis (PVT) have been controversial. In this study the investigators wanted to identify the most effective and safe regimen among different thrombolytic strategies.Transesophageal echocardiography (TEE) guided thrombolytic treatment was administered to 182 consecutive patients with PVT in 220 different episodes (156 women, mean age 43.2±13.06 years) between 1993 and 2009. These regimens included rapid streptokinase (Group I, 16 episodes), slow streptokinase (Group II, 41 episodes), high dose (100 mg) tissue plasminogen activator (t-PA) (Group III, 12 episodes), half-dose (50 mg) slow infusion (6-hours) of t-PA without bolus (Group IV, 27 episodes), and low dose (25 mg) and slow infusion (6-hours) of t-PA without bolus (Group V, 124 episodes). The study endpoints were thrombolytic success and in-hospital mortality and non-fatal complication rates.

DETAILED DESCRIPTION:
One hundred and eighty two consecutive in-hospital patients with 220 episodes of PVT between 1993 and 2009 were included in the study. The patients were enrolled after informed consent if there was no contraindication, to thrombolysis. The study was approved by the local Ethics Board. The patient demographics, past medical history, date of the operation, type and make of the prosthetic valve, rhythm disorders, aspirin use, NYHA functional capacity, leading symptoms and international normalization ratio (INR) values at the time of admission were prospectively entered into a database.The diagnosis of PVT was verified each time by transesophageal echocardiography (TEE) when a patient was admitted with thromboembolism or persistently low INR for the preceding consecutive 3 months and when a transthoracic echocardiography (TTE) documented prosthetic valve dysfunction or thrombus. All patients underwent TTE and TEE examination before and after the thrombolysis sessions. The cross sectional area and the longest diameter of the thrombus were measured on TEE recordings

ELIGIBILITY:
Inclusion Criteria:

* Patients with prosthetic valve thrombosis

Exclusion Criteria:

* Large left atrial thrombus
* Recent (<3 weeks) ischemic stroke
* Hemorrhagic stroke
* Early (<4 days) postoperative period
* Traumatic accident <4 weeks
* Bleeding diathesis †
* İntracranial mass
* Active internal bleed
* Aortic dissection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 1993-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Thrombolytic success | 24 hours
  In the absence of fatal or nonfatal major complications;
  * Obstructive thrombus:
    1. Doppler documentation of the resolution of increased gradient and decreased valve area.
    2. Clinical improvement in symptoms.
    3. Reduction by ≥75% in major diameter or area of the thrombus. Complete success was defined when all 3 criteria were met and partial success was defined as less than 3.
  * Nonobstrucive thrombus:
    1. Complete success: ≥75% reduction in thrombus area.
    2. Partial success: 50%-75% reduction in thrombus area.
Non-fatal complication rates | participants will be followed for the duration of hospital stay, an expected average of 3 weeks
  * Nonfatal major complication: Ischemic stroke, intracranial hemorrhage, embolism (coronary or peripheral), bleeding requiring transfusion.
  * Nonfatal minor complication: Bleeding without need for transfusion, TIA.
In-hospital mortality | participants will be followed for the duration of hospital stay, an expected average of 3 weeks
  All cause in-hospital mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Ozkan, Assoc.Prof., Principal Investigator — Kosuyolu Kartal Heart Training and Research Hospital
Locations (1):
- Kosuyolu Kartal Heart Training and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Ozkan M, Kaymaz C, Kirma C, Sonmez K, Ozdemir N, Balkanay M, Yakut C, Deligonul U. Intravenous thrombolytic treatment of mechanical prosthetic valve thrombosis: a study using serial transesophageal echocardiography. J Am Coll Cardiol. 2000 Jun;35(7):1881-9. doi: 10.1016/s0735-1097(00)00654-9. PMID 10841239
- [Derived] Ozkan M, Gunduz S, Biteker M, Astarcioglu MA, Cevik C, Kaynak E, Yildiz M, Oguz E, Aykan AC, Erturk E, Karavelioglu Y, Gokdeniz T, Kaya H, Gursoy OM, Cakal B, Karakoyun S, Duran N, Ozdemir N. Comparison of different TEE-guided thrombolytic regimens for prosthetic valve thrombosis: the TROIA trial. JACC Cardiovasc Imaging. 2013 Feb;6(2):206-16. doi: 10.1016/j.jcmg.2012.10.016. PMID 23489534